HIC#: 2000023271

# CONSENT FOR PARTICIPATION IN A RESEARCH PROJECT YALE UNIVERSITY SCHOOL OF MEDICINE – YALE-NEW HAVEN HOSPITAL

200 FR. 7 (2016-1)

Study Title: Preventing Childhood Obesity Through a Mindfulness-Based Parent Stress

Intervention

Principal Investigator: Rajita Sinha PhD

Funding Source: National Institute of Diabetes and Digestive and Kidney Diseases/NIH/DHHS

## **ADDENDUM**

This consent addendum gives new information about the research study in which you agreed to participate. Your study research staff member will discuss this new information with you. The new questionnaire noted below is in addition to those which you were informed about in the previous consent form. You should know enough about this study's risks and benefits to make an informed judgment about whether or not you wish to continue to take part in the research. Once you understand the new information, you will be asked to sign this form. This process is known as informed consent. You will receive a copy of this signed form for your records.

## **Brief Description of the Project**

The purpose of the study you previously participated in and completed is to learn about stress, diet, and exercise. It is our belief that the results of our study may make it possible for us to better understand the role of family stress and healthy choices in the development of children. As part of your agreement to take part in this study, you have been asked to participate in intake appointments, blood work, the toy-wait task, and a 12-week group, as well as 4 follow up appointments over a 2 year period. You may have also attend a number of these appointments and attend the groups via the internet or phone if needed.

### **New Risks, Additional Information**

There are no new risks associated with this study.

#### **New Procedure(s)**

If you agree to continue your participation in this study, you will be asked to complete one brief follow up phone survey regarding your weight and health history since participating in the study. The phone survey should take around 5 minutes to complete. You will be compensated with a \$10 gift card for completing this survey.

| □ I willingly co | sent to participate in the study-specific follow up survey | 7. |
|---|---|---|
| Initials: | Date: | |
| Version #1 | Page 1 of 2 | |

#### APPROVED BY THE YALE UNIVERSITY IRB 7/5/2022

HIC#: 2000023271

| ☐ I do not wish to participate in the study-sp | pecific follow up survey. |
|---|---|
| Initials:Date: | |
| Authorization I have read (or someone has read to me) this form the project described above. Its general purposes hazards and inconveniences have been explained that I have received a copy of this consent addended. | s, the particulars of involvement and possible to my satisfaction. My signature also indicates |
| Name of Subject: | - |
| Signature: | - |
| Date: | |
| Signature of Person Obtaining Consent | Date |

If you have further questions about this project or if you have a research-related problem, you may contact the Principal Investigator (Dr. Rajita Sinha 203-737-5805). If you would like to talk with someone other than the researchers to discuss problems, concerns, and questions, offer input, discuss situations in the event that a member of the research team is not available, or if you have any questions concerning your rights as a research subject, you may contact the Human Investigation Committee at (203) 785-4688.